CLINICAL TRIAL: NCT00815607
Title: Phase 1b' Open Label, Single Arm, Multicenter Trial to Evaluate the Safety, Tolerance, Response Rate and Immunological Effects of Repeated Intratumoral Injections of Adenoviral Transduced Autologous Dendritic Cells Engineered to Express hIL-12(INXN-3001) in Response to an Oral Activator Ligand in Patients With Unresectable Stage III C or IV Malignant Melanoma
Brief Title: Trial of an Intratumoral Injections of INXN-3001 in Subjects With Stage III or IV Melanoma
Status: Completed | Phase: Phase 1 | Type: Interventional
Sponsor: Alaunos Therapeutics (Industry)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: RTS-M101B'; NIH OBA 0710-881
Record Dates: First submitted 2008-12-19; First posted 2008-12-30 (Estimated); Last update posted 2013-07-18 (Estimated); Status verified 2013-07

CONDITIONS: Melanoma
Keywords: melanoma; biologic; immunotherapy; cancer
MeSH Terms: conditions — Melanoma; Neoplasms

INTERVENTIONS:
Drug: INXN-1001 — Capsules given once daily for 14 days for 3 treatment cycles.
Biological: INXN-3001 — Intratumoral injection

SUMMARY:
The purpose of this study is to test the safety of an investigational combination drug/immunotherapy for the treatment of Stage III/IV melanoma.

DETAILED DESCRIPTION:
This study will examine the effects of an oral Activator Ligand administration to modulate the timing of gene expression of human IL-12 by adenovirus-transduced dendritic cells injected into tumors.

ELIGIBILITY:
Inclusion Criteria:

1. Males or females of all races ≥ 18 years of age and ≤ 75 years of age;
2. Unresectable Stage III C (in transit) or Stage IV melanoma (M1a, M1b, M1c with LDH ≤ 2x ULN), arising from primary cutaneous, mucosal, or subungual melanoma of any tumor thickness or from an unknown primary site;
3. A minimum of 2-3 accessible nonvisceral lesions (longest diameter ≤3 cm) or palpable tumor-involved lymph nodes (longest diameter ≤5 cm) for intratumoral injections (INXN-3001) and biopsies;
4. ECOG performance status of 0 or 1;
5. Patients without visible brain metastases as assessed by contrast-enhanced MRI scan within 6 weeks prior to receiving study treatment;
6. Adequate baseline hematological and organ function, assessed by laboratory values within 42 days (6 weeks) prior to study entry and prior to repeat treatment cycles with INXN-1001 as follows: hemoglobin ≥ 10 g/L, granulocytes > 2500/mm3, lymphocytes > 1000/ mm3, platelets > 100,000/ mm3, serum creatinine < 1.5 x ULN, AST, ALT, alkaline phosphatase < 2.5 x ULN, LDH ≤ 2 x ULN, serum bilirubin < 1.5 x ULN, absolute neutrophils > 500/ mm3;
7. An expected survival of at least approximately 6 months in the opinion of the investigator (as assessed mainly by performance status);
8. Females must be post-menopausal or surgically sterile or practice effective contraception; Men who are not surgically sterile and whose partners are not post-menopausal or surgically sterile must practice effective contraception;
9. Normal coagulation parameters as measured by PT/PTT;
10. Signed, IRB-approved voluntary written informed consent.

Exclusion Criteria:

1. Active, acute viral, bacterial, or fungal infections requiring specific therapy;
2. HIV-infection due to concerns about ability to mount an effective immune response;
3. Active autoimmune disease requiring steroids (>10 mg prednisolone or comparable) or other immunosuppressive therapy;
4. Patients with detectable brain metastases at the time of screening (or within 6 weeks prior to receiving study treatment), as assessed by contrast-enhanced MRI scans;
5. Patients with one or more lesion(s) > 3cm (LD) or palpable, tumor-involved lymph node(s) >5 cm (LD);
6. Patients with a hemoglobin of < 10 g/L;
7. Presence of Stage IV visceral metastases or other distant metastases if LDH >2 x ULN;
8. Patients who have previously been treated with INXN-3001 and INXN-1001;
9. Recipients of organ allografts;
10. Other concurrent, clinically active malignant disease, with the exception of other cancers of the skin;
11. Less than 30 days (before the first dose of study medication) have elapsed since the completion of prior chemotherapy, hormonal therapy, radiotherapy, immunotherapy, or any first line therapy;
12. Clinically significant cerebrovascular disease;
13. History of or concurrent severe cardiac insufficiency (New York Heart Association Class III or IV) or coronary artery disease;
14. QTc interval of >470 ms on screening;
15. Inability to measure the QT interval due to conduction abnormalities such as Bundle Branch Block (left or right) or persistent cardiac arrhythmia e.g. atrial fibrillation, or cardiac pacemaker;
16. Long QT syndrome or family history of sudden cardiac death in young family members;
17. Concomitant use of medication known to affect ventricular repolarization;
18. Cardiac comorbidity such as a left ventricular ejection fraction <45%, myocardial infarction, persistent angina, or cardiac surgery within 3 months prior to enrollment;
19. Uncontrollable hypertension (>150 mm Hg systolic or >100 mm Hg diastolic);
20. Acute medical conditions such as ischemic heart or lung disease that may be considered an unacceptable anesthetic or operative risk;
21. History of or current bleeding or uncorrected clotting disorders;
22. Concurrent immunosuppressive therapy such as corticosteroids (>10mg prednisolone or comparable) and cyclosporin A;
23. Concurrent investigational treatments, or treatment with any investigational treatment within the past 30 days (prior to the first dose of study medication);
24. Concurrent medications that are metabolized by the CYP 3A4 pathway;
25. Females who are lactating or pregnant;
26. A Body Mass Index (BMI) greater than or equal to 40 kg/m2; aa. Patients who have a history of hypersensitivity that may relate to any component of the product, e.g. to benzoic acid that might be related to INXN-1001, which contains two benzene rings; bb. Any medical or psychiatric condition which, in the opinion of the investigator, would unacceptably reduce the safety or delivery of the proposed treatment, or would preclude obtaining voluntary informed consent.

Ages: 18 Years to 75 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 12 (Actual)
Dates: Start 2009-04; Primary Completion 2013-01 (Actual); Study Completion 2013-01 (Actual)

PRIMARY OUTCOMES:
Physical examinations, vital signs, serum chemistry, urinalysis, hematology, adverse events, and objective response rate, as assessed by diagnostic CT scans | throughout the study

SECONDARY OUTCOMES:
PK of oral Activator Ligand, Immunologic responses, particularly frequency of CTLs and Tregs and hIL-12 and other cytokine levels in injected target tumor(s) and in peripheral blood, Efficacy. | throughout the study

CONTACTS AND LOCATIONS:
Overall Officials: Andrew Marsh, Study Director — Ziopharm Oncology
Locations (8):
- United States (8):
  - The Angeles Clinic and Research Institute, Santa Monica, California
  - Helen F. Graham Cancer Center, Newark, Delaware
  - • Nancy N. and J.C. Lewis Cancer Center & Research Pavilion at St. Joseph/Candles, Savannah, Georgia
  - Oncology Specialists, S.C., Park Ridge, Illinois
  - Goshen Clinic, Goshen, Indiana
  - Billings Clinic, Billings, Montana
  - Penn State Milton S. Hershey Medical Center, Hershey, Pennsylvania
  - Mary Crowley Cancer Research Centers, Dallas, Texas